CLINICAL TRIAL: NCT02882295
Title: Validation of the Zigzag Tracking Task Test for the Evaluation of Handwriting Difficulties in Writer's Cramp
Acronym: LabyDys
Status: Terminated | Type: Observational
Why Stopped: recrutement difficulties
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SSA_2016_10
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Dystonic Disorder
MeSH Terms: conditions — Dystonic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- writer's cramp: patients assessed without, then with Botulinum Neurotoxin injections
  Interventions: Other: Validation of a handwriting scale
- control: age and gender matched
  Interventions: Other: Validation of a handwriting scale

INTERVENTIONS:
Other: Validation of a handwriting scale

SUMMARY:
Writer's cramp (WC) is a task specific dystonia that occurs from the moment patient starts writing. It leads to partial or complete inability to use the hand only during the handwriting gesture. It is characterized by the appearance of cramps or spasms of certain muscles of the hand and/or forearm.

Clinical scales currently use for the assessment of WC fail to accurately reflect changes in the characteristics of handwriting in response to treatments (Botulinum Neurotoxin injections and / or retraining therapy).

The Zigzag Tracking Task (ZZTT), easy to use in current practice provides useful information in terms of speed and precision of handwriting gesture. This timed handwriting test is to follow with a pen a zigzag path beset with obstacles to avoid. It permits to evaluate the time in seconds required to carry out the zigzag path and count the number of errors (output path and contacts with obstacles). The investigators propose to validate the ZZTT for the assessment of the handwriting gesture of WC.

ELIGIBILITY:
Inclusion Criteria:

* scholarship in French language, at least until 16 years old
* writer's cramp (diagnostic confirmed by a neurologist specialized in movement disorders)
* prescription of botulinum neurotoxin injection
* prescription de novo or absence of injection in the last 3 months
* informed consent
* medical insurance coverage

Exclusion Criteria:

* writing tremor
* -other neurological disease with effect on handwriting
* pain or traumatism of the upper limb, with effect on handwriting
* non-corrected visual disturbances
* patient living outside the region where the study will be held (Ile-de-France)
* participation in another research with a potential impact on evaluation criteria
* pregnant or breast feeding patient
* patient under judiciary protection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients suffering from writer's cramp and healthy subjects, age and gender matched
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
hand-writing speed | immediate
  speed and accuracy of handwriting

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BLETON, PhD, Study Director — Fondation OPH A de Rothschild; Sophie SANGLA, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France